CLINICAL TRIAL: NCT03348462
Title: Formulation and Clinical Evaluation of Ethosomal and Liposomal Preparations of Anthralin in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Kamal, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: faceoealpoaip
Record Dates: First submitted 2017-10-30; First posted 2017-11-21 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Psoriasis Vulgaris
Keywords: psoriasis; anthralin; ethosome; liposome
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: The aim of the present study was to develop an ethosomal delivery system anthralin and evaluate its effectiveness and safety in treatment of psoriasis and comparing it with liposomal delivery system anthralin.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ethosomal anthralin (Experimental): Group 1: included 10 psoriatic patients will be treated with ethosomal preparation of anthralin. Patients will be treated with this preparation with short contact (only one hour) daily up to 8 weeks.
  Interventions: Drug: ethosomal preparation of anthralin
- liposomal anthralin (Active Comparator): Group 2: included 10 psoriatic patients will be treated with liposomal preparation of anthralin. Patients will be treated with this preparation with short contact (only one hour) daily up to 8 weeks.
  Interventions: Drug: liposomal preparation of anthralin

INTERVENTIONS:
Drug: ethosomal preparation of anthralin — once daily with short contact topical application
  Arms: ethosomal anthralin
Drug: liposomal preparation of anthralin — once daily with short contact topical application
  Arms: liposomal anthralin

SUMMARY:
Psoriasis is a common immune mediated inflammatory skin disease characterized by red heavily scaled plaques. Anthralin (1,8-dihydroxy-9-anthrone) which was introduced over 80 years ago has shown excellent efficacy in the management of psoriasis.Although anthralin is remarkably effective in the management of psoriasis, its side effects are equally disturbing. Its use is messy as it stains the skin, clothing, and any furniture that it may come in contact with. Further, anthralin has irritating, burning, brown discoloration and necrotizing effect on the normal and the diseased skin. This troublesome profile has discouraged wide-spread use of the drug.

Ethosomes are attractive vesicular carriers mainly composed of phospholipids, ethanol and water. The intriguing features of ethosomes are due to their high ethanol content which facilitate their penetration through stratum corneum and target deep skin layers. This is advantageous over conventional liposomes which have limited penetration through the skin and remain confined in the upper layer of the stratum corneum. Compared to liposomes, ethosomes had greater retention of methotrexate into the skin for a longer period of time, suggesting better therapeutic outcome.

DETAILED DESCRIPTION:
Psoriasis is a common immune mediated inflammatory skin disease characterized by red heavily scaled plaques. Anthralin (1,8-dihydroxy-9-anthrone) which was introduced over 80 years ago has shown excellent efficacy in the management of psoriasis.Anthralin mechanism of action involves inhibition of the proliferation of keratinocytes. Further, accumulation of anthralin inside the mitochondria impairs energy supply to the cell, probably due to the free radicals resulting from oxidation of the drug. Anthralin also interferes with the replication of DNA and slows down the extreme cell division that occurs in psoriatic plaques. Although anthralin is remarkably effective in the management of psoriasis, its side effects are equally disturbing. Its use is messy as it stains the skin, clothing, and any furniture that it may come in contact with. Further, anthralin has irritating, burning, brown discoloration and necrotizing effect on the normal and the diseased skin. This troublesome profile has discouraged wide-spread use of the drug.

Ethosomes are attractive vesicular carriers mainly composed of phospholipids, ethanol and water. The intriguing features of ethosomes are due to their high ethanol content which facilitate their penetration through stratum corneum and target deep skin layers. This is advantageous over conventional liposomes which have limited penetration through the skin and remain confined in the upper layer of the stratum corneum. Compared to liposomes, ethosomes had greater retention of methotrexate into the skin for a longer period of time, suggesting better therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients with mild to moderate, stable chronic plaque psoriasis.

Exclusion Criteria:

* patients with severe psoriasis.
* Patients received any topical or systemic treatment for psoriasis one month before the start of the study.

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) score | up to 8 weeks
  PASI combines the assessment of the severity of psoriatic lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). PASI will be measured before and after treatment to assess the efficacy of therapy.Steps in generating PASI score
  1. Divide body into four areas: head, arms, trunk, and legs .
  2. Generate an average score for the erythema, thickness, and scaling for each of the 4 areas , each graded on a 0-4 scale (0 = clear, 1= slight,2= mild, 3=moderate, 4=severe).
  3. Sum scores of erythema, thickness, and scale for each area.
  4. Generate a percentage for skin covered with psoriasis for each area and convert that to a 0-6 scale (0 = 0%; 1 =,10%; 2 = 10-,30%; 3 = 30-,50%; 4 = 50-
     ,70%; 5 = 70-,90%; 6 = 90-100%).
  5. Multiply score of item (c) above times item (d) above for each area and multiply that by 0.1, 0.2, 0.3, and 0.4 for head, arms, trunk, and legs, respectively.
  6. Add these scores to get the PASI score.

SECONDARY OUTCOMES:
Histopathological examination of psoriatic lesions using hematoxylin and eosin staining (H & E stain) | up to 8 weeks
  hematoxylin and eosin staining of skin biopsies from psoriatic lesions before and after treatment will be done.
Safety of the drug perparations | up to 8 weeks
  by recording any possible adverse events like itching, burning sensation, staining of skin or clothes and erythema.
Patient satisfaction | up to 8 weeks
  at the end of treatment, it will be evaluated by patient's self assessment of the degree of improvement of psoriasis
digital photography | up to 8 weeks
  digital photography of the lesions before and after treatment using a 14.1 megapixels Sony DSC- W 390 digital camera will be done for each patient to assess any changes in clinical appearance of psoriatic lesions and evaluate the response of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Hollywood KA, Winder CL, Dunn WB, Xu Y, Broadhurst D, Griffiths CE, Goodacre R. Exploring the mode of action of dithranol therapy for psoriasis: a metabolomic analysis using HaCaT cells. Mol Biosyst. 2015 Aug;11(8):2198-209. doi: 10.1039/c4mb00739e. PMID 26018604
- [Background] Parish LC, Millikan LE, Witkowski JA. The modern story of anthralin. Int J Dermatol. 1989 Jul-Aug;28(6):373-4. doi: 10.1111/j.1365-4362.1989.tb02481.x. No abstract available. PMID 2767834
- [Background] Saraswat A, Agarwal R, Katare OP, Kaur I, Kumar B. A randomized, double-blind, vehicle-controlled study of a novel liposomal dithranol formulation in psoriasis. J Dermatolog Treat. 2007;18(1):40-5. doi: 10.1080/09546630601028729. PMID 17365266
- [Background] McGill A, Frank A, Emmett N, Turnbull DM, Birch-Machin MA, Reynolds NJ. The anti-psoriatic drug anthralin accumulates in keratinocyte mitochondria, dissipates mitochondrial membrane potential, and induces apoptosis through a pathway dependent on respiratory competent mitochondria. FASEB J. 2005 Jun;19(8):1012-4. doi: 10.1096/fj.04-2664fje. Epub 2005 Mar 31. PMID 15802490
- [Background] Mendonca CO, Burden AD. Current concepts in psoriasis and its treatment. Pharmacol Ther. 2003 Aug;99(2):133-47. doi: 10.1016/s0163-7258(03)00041-x. PMID 12888109
- [Background] Sehgal VN, Verma P, Khurana A. Anthralin/dithranol in dermatology. Int J Dermatol. 2014 Oct;53(10):e449-60. doi: 10.1111/j.1365-4632.2012.05611.x. Epub 2014 Sep 10. PMID 25208745
- [Background] Agarwal R, Katare OP, Vyas SP. Preparation and in vitro evaluation of liposomal/niosomal delivery systems for antipsoriatic drug dithranol. Int J Pharm. 2001 Oct 9;228(1-2):43-52. doi: 10.1016/s0378-5173(01)00810-9. PMID 11576767
- [Background] Pradhan M, Singh D, Singh MR. Novel colloidal carriers for psoriasis: current issues, mechanistic insight and novel delivery approaches. J Control Release. 2013 Sep 28;170(3):380-95. doi: 10.1016/j.jconrel.2013.05.020. Epub 2013 Jun 13. PMID 23770117
- [Background] Dubey V, Mishra D, Dutta T, Nahar M, Saraf DK, Jain NK. Dermal and transdermal delivery of an anti-psoriatic agent via ethanolic liposomes. J Control Release. 2007 Nov 6;123(2):148-54. doi: 10.1016/j.jconrel.2007.08.005. Epub 2007 Aug 16. PMID 17884226
- [Background] Touitou E, Dayan N, Bergelson L, Godin B, Eliaz M. Ethosomes - novel vesicular carriers for enhanced delivery: characterization and skin penetration properties. J Control Release. 2000 Apr 3;65(3):403-18. doi: 10.1016/s0168-3659(99)00222-9. PMID 10699298
- [Derived] Fathalla D, Youssef EMK, Soliman GM. Liposomal and Ethosomal Gels for the Topical Delivery of Anthralin: Preparation, Comparative Evaluation and Clinical Assessment in Psoriatic Patients. Pharmaceutics. 2020 May 11;12(5):446. doi: 10.3390/pharmaceutics12050446. PMID 32403379
- See also: Nanotechnology in dermatology — http://www.biomedsearch.com/nih/Nanotechnology-in-dermatology/24626657.html